CLINICAL TRIAL: NCT02997397
Title: A Novel Atraumatic Tourniquet Technique in Cases of Excessive Bleeding During Cesarean Section
Brief Title: A Novel Tourniquet Technic for Massive PPH
Acronym: PPH
Status: Completed | Type: Observational
Sponsor: Irenbe (Other)
Responsible Party: Principal Investigator, Baris Buke, M.D., Irenbe
Other Study IDs: IR-2016-01
Record Dates: First submitted 2016-12-10; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tourniquets

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- tourniquet (+): The cases in which the tourniquet technique is used
  Interventions: Procedure: tourniquet(+)
- tourniquet(-): The cases in which the tourniquet technique is not used
  Interventions: Procedure: tourniquet(-)

INTERVENTIONS:
Procedure: tourniquet(+) — A novel atraumatic tourniquet technique, applied via placing a vascular clamp widely on both the infundibulopelvic ligament and uterine arteries.
  Groups: tourniquet (+)
Procedure: tourniquet(-)
  Other Names: The tourniquet was not used
  Groups: tourniquet(-)

SUMMARY:
In this study, the investigators aimed to find out the effect of a novel tourniquet technique, in cases of excessive bleeding during cesarean delivery.

DETAILED DESCRIPTION:
In this retrospective comparative study, the investigators compared the peripartum features of patients who experienced profuse postpartum bleeding during C/S and this novel atraumatic tourniquet technique was used and not used.

In this technique; the uterus is exteriorized following the delivery of the baby and before the removal of the placenta to be able to apply the tourniquet technique. In this technique it is not obligatory to push the bladder before the procedure. Afterwards, the surgeon and the assistant palpate the ureters with both hands in the two sheaths of broad ligament and try to hear a 'click' sound which comes from ureter sliding out between both fingers. After confirming that the ureters are not in the surgical site, an atraumatic vascular DeBakey clamp is applied widely including both the infundibulopelvic ligament and uterine arteries. Thus, two-sided blood supply of the uterus is reduced significantly and this gives the surgeon some time, for planning further surgical procedures and also serves a minimal bloody surgical site. If the avascular state of the surgical site is needed for a prolonged time, for instance while preparing for a blood transfusion or while waiting until an experienced surgeon is available, the clamps were opened and closed intermittently for a maximum of 10 minutes, as to sustain the blood supply of the ovaries and the uterus.

ELIGIBILITY:
Inclusion Criteria:

* The women who experienced profuse postpartum haemorrhage during cesarean section

Exclusion Criteria:

* none defined

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Two groups of women who experienced profuse bleeding during C/S; one group in which a novel tourniquet technique was used and another group in which the tourniquet technique was not used.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Hemoglobin values | 1 hour
  The differences in hemoglobin values just before the surgery and immediately after the surgery
red blood cell transfusion | 24 hours
  the amount of packed red blood cells, required for haemodynamic stability in the first 24 hour.
fresh frozen plasma transfusion | 24 hours
  the amount of packed fresh frozen plasma, required for haemodynamic stability in the first 24 hour.

CONTACTS AND LOCATIONS:
Overall Officials: Barış Büke, resident, Principal Investigator — İRENBE
Locations (1):
- Ege University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If needed

REFERENCES:
- [Result] B-Lynch C, Coker A, Lawal AH, Abu J, Cowen MJ. The B-Lynch surgical technique for the control of massive postpartum haemorrhage: an alternative to hysterectomy? Five cases reported. Br J Obstet Gynaecol. 1997 Mar;104(3):372-5. doi: 10.1111/j.1471-0528.1997.tb11471.x. PMID 9091019
- [Result] Hayman RG, Arulkumaran S, Steer PJ. Uterine compression sutures: surgical management of postpartum hemorrhage. Obstet Gynecol. 2002 Mar;99(3):502-6. doi: 10.1016/s0029-7844(01)01643-x. PMID 11864681
- [Result] AbdRabbo SA. Stepwise uterine devascularization: a novel technique for management of uncontrolled postpartum hemorrhage with preservation of the uterus. Am J Obstet Gynecol. 1994 Sep;171(3):694-700. doi: 10.1016/0002-9378(94)90084-1. PMID 8092217
- [Result] Ikeda T, Sameshima H, Kawaguchi H, Yamauchi N, Ikenoue T. Tourniquet technique prevents profuse blood loss in placenta accreta cesarean section. J Obstet Gynaecol Res. 2005 Feb;31(1):27-31. doi: 10.1111/j.1447-0756.2005.00247.x. PMID 15669988